CLINICAL TRIAL: NCT03250468
Title: Sleep to Your Heart's Content - Insomnia Intervention for Cardiac Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor follow/up rates and data.
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Heather Tulloch, Clinical Psychologist, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6997
Record Dates: First submitted 2017-07-27; First posted 2017-08-15 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Insomnia; Cardiovascular Diseases
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-I (Experimental): Participants randomized to receive the intervention will attend 6 weekly group-based CBT-I sessions. Each 90-minute group will include 6-12 participants.
  Interventions: Behavioral: CBT-I
- Wait-list control (No Intervention): The wait-list control group will receive treatment as per our standard cardiac rehabilitation program. After completion of the 3-month follow-up questionnaire, wait-list control participants may take part in the intervention.

INTERVENTIONS:
Behavioral: CBT-I — Each weekly session will focus on several psychological and behavioural techniques that include sleep restriction, relaxation strategies, cognitive therapy, stimulus control therapy, and education about proper sleep hygiene.
  Arms: CBT-I

SUMMARY:
Research aims:

1. To determine if participation in a group-based cognitive behavioural therapy intervention (CBT-I) intervention results in improved sleep quality.
2. To determine if participation in a group-based CBT-I intervention results in improved cardiovascular disease risk factors, and if the CBT-I intervention moderates that relationship.

DETAILED DESCRIPTION:
Cardiovascular disease affects 5% of the population and almost 20% of those meet the criteria for insomnia; twice as many as in the general population. Patients with cardiovascular disease and insomnia have been found to have elevated rates of anxiety and depression, which in turn places individuals at further cardiovascular risk via physiological pathways like increased blood pressure and/or vascular inflammation. Further, insomnia has been linked with negative health outcomes that exacerbate risk, including obesity, hypertension, and future acute myocardial infarction. Given the negative impact of poor sleep on cardiac health, some have argued that insomnia should now be included in the top 10 modifiable risk factors for cardiovascular disease.

Currently the best treatment for insomnia is a group-based cognitive behavioural therapy intervention (CBT-I); this intervention is more effective than pharmacotherapy. Evidence shows that CBT-I produces significant improvements after 6 weeks of intervention and improvements continue over the long term. This intervention program includes specific cognitive therapy exercises aimed at maladaptive thoughts about sleep, behaviour change techniques, and relaxation strategies (e.g., mindfulness, deep breathing); it also provides a supportive environment for individuals to discuss their sleep difficulties, allowing them to feel normalized and less isolated. For most people with insomnia however, their disorder goes untreated, leaving individuals at higher risk for affective disorders (e.g., depression), cardiovascular disease, and poorer quality of life. This lack of treatment is widespread and systemic; patients who want help with insomnia face a dearth of information about treatment, actual access to treatment and affordable services.

The proposed study is the first evaluation of a comprehensive CBT-I intervention designed for cardiac patients. Of note, the proposed study will be the first to evaluate the impact of this intervention on cardiovascular outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Sleep disturbance as indicated by a score on the Insomnia Severity Index (ISI) of 8 or above.
* Enrolled in the cardiac rehabilitation program offered by the University of Ottawa Heart Institute.
* Willing to be randomized.
* Willing to wear a monitor that tracks sleep and physical activity.

Exclusion Criteria:

* Untreated or undiagnosed obstructive sleep apnea (as per standard cardiac rehabilitation intake assessment, patients with a score of 5 or above on the STOP-BANG (a brief assessment for sleep apnea) will be referred for a sleep assessment by a cardiac rehabilitation physician).
* Unable to converse in English (i.e., while patient materials and questionnaires will be offered in both English and French, the intervention is only offered in English).
* Unable to provide written, informed consent.
* Unable to attend 6 weeks of onsite CBT-I intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | Through study completion, up to 3 months
  Sleep quality will be measured using the Consensus Sleep Diary.

SECONDARY OUTCOMES:
Sleep Symptoms | Through study completion, up to 3 months
  Sleep symptoms will be measured using the Insomnia Severity Index
Sleepiness | Through study completion, up to 3 months
  The widely used Epworth Sleepiness Scale will be used to measure levels of sleepiness .experienced by patients
Activity | Through study completion, up to 3 months
  Participants will wear an ActiGraph GTX3 accelerometer (ActiGraph, Pensacola, Florida) to assess sleep and physical activity
Mental Health | Through study completion, up to 3 months
  Both symptoms and severity of anxiety and depression will be measured
Quality of life | Through study completion, up to 3 months
  Patient quality of life will be measured using the 36-item short-form health survey (SF-36; version 1)
Cardiovascular Risk Factors | Through study completion, up to 3 months
  Cardiovascular disease diagnosis, fasting blood glucose concentration, triglycerides, glycated hemoglobin (HbA1c), cholesterol (High-density lipoprotein ratio

CONTACTS AND LOCATIONS:
Overall Officials: Heather Tulloch, Ph.D, Principal Investigator — Clinical, Health, and Rehabilitation Psychologist
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada